CLINICAL TRIAL: NCT04029090
Title: A Randomized, Single-Blind, Placebo-Controlled, Three-Way Crossover Study to Evaluate the Effect of MCI-186 at Therapeutic and Supra-Therapeutic Doses on the QT/QTc Interval in Healthy Subjects
Brief Title: A Study to Evaluate the Effect of MCI-186 at Therapeutic and Supra-Therapeutic Doses on the QT Interval(QT)/Corrected QT Interval(QTc) Interval in Healthy Subjects
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Tanabe Pharma Corporation (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Other
Other Study IDs: MCI-186-J25
Record Dates: First submitted 2019-07-10; First posted 2019-07-23 (Actual); Results first posted 2024-11-21 (Actual); Last update posted 2026-01-08 (Actual); Status verified 2025-12

CONDITIONS: Healthy Adult Subjects
MeSH Terms: interventions — Edaravone

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Masking Description: This study is a single-blind study. Subjects and Electrocardiogram (ECG) reviewer will be blinded. Investigator and Sponsor will be unblinded.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- Sequence 1 (Experimental): Subjects will receive a single intravenous dose of MCI-186 as a 1-hour infusion in the treatment sequence: first Treatment A, then Treatment C, then Treatment B (Treatment A= 60 mg of MCI-186, Treatment B= 300 mg of MCI-186, treatment C=0.9% w/v saline)
  Interventions: Drug: MCI-186; Drug: Placebo
- Sequence 2 (Experimental): Subjects will receive a single intravenous dose of MCI-186 as a 1-hour infusion in the treatment sequence: first Treatment B, then Treatment A, then Treatment C (Treatment A= 60 mg of MCI-186, Treatment B= 300 mg of MCI-186, treatment C=0.9% w/v saline)
  Interventions: Drug: MCI-186; Drug: Placebo
- Sequence 3 (Experimental): Subjects will receive a single intravenous dose of MCI-186 as a 1-hour infusion in the treatment sequence: first Treatment C, then Treatment B, then Treatment A (Treatment A= 60 mg of MCI-186, Treatment B= 300 mg of MCI-186, treatment C=0.9% w/v saline)
  Interventions: Drug: MCI-186; Drug: Placebo

INTERVENTIONS:
Drug: MCI-186 — A single dose of 60 mg MCI-186 over 60 min will be intravenously administered.
  Other Names: Edaravone
Drug: MCI-186 — A single dose of 300 mg MCI-186 over 60 min will be intravenously administered.
  Other Names: Edaravone
Drug: Placebo — A single dose of 0.9% w/v saline over 60 min will be intravenously administered.

SUMMARY:
To evaluate the effect of MCI-186 on the QT interval corrected for heart rate using Fridericia's formula (QTcF)

ELIGIBILITY:
Inclusion Criteria:

* Healthy males aged 20 to 55 years (both inclusive) at signature of the Informed Consent Form (ICF).
* Able to provide written informed consent to participate in this study after reading the ICF, and after having the opportunity to discuss the study with the Investigator or designee, before any screening or study related procedures take place.
* In the Investigator's opinion, subject is able to understand the nature of the study and any risks involved in participation, and willing to cooperate and comply with the protocol restrictions and requirements.
* A body weight of ≥45 kg and a body mass index (BMI) ranging from 18 to 30 kg/m2 (both inclusive) at screening and Day -1.
* Good health and free from clinically significant illness or disease in the opinion of the investigator on the basis of a physical examination, medical history, ECG, vital sign, and clinical laboratory test (biochemistry, hematology, coagulation and urinalysis) at screening and Day -1.
* Male subjects must practice effective contraception during the study, from the time of the first dose of Investigational Medicinal Product (IMP) until 14 days after the last dose of IMP.

Exclusion Criteria:

* Subjects with PR >240 msec, QRS ≥120 msec, or QTcF >450 msec on the screening or Day -1 ECG, or any clinically significant electrocardiographic abnormality in the opinion of the Investigator.
* Subject who has a history of cardiac disease or arrhythmias that can cause QTc prolongation.
* Subject who has a family history of Torsade de Pointes, long-QT syndrome, hypokalemia or sudden death.
* Subjects with potassium levels outside of the laboratory reference ranges at screening or Day -1.
* Subjects with clinically significant deviations from normal in physical examination, vital signs, ECG or clinical laboratory test at screening or Day -1 in the opinion of the Investigator.
* Presence or history of any clinically significant disease or organ dysfunction in the opinion of the Investigator.
* Presence or history of allergy to food, any medical product or relevant excipient that is of clinical significant.
* Subjects were previously administered MCI-186.
* Presence or history of alcohol abuse or a positive alcohol test.
* Presence or history of drug abuse or a positive drug screen test.
* Positive test for hepatitis C virus antibody, hepatitis B surface antigen, human immunodeficiency virus (HIV) antigen/antibody or syphilis test at screening.
* Participation in another trial within 12 weeks or 5 times the half-life of the drug whichever is longer before providing a signed ICF. For biologics, the minimum period is at least 24 weeks or the period of the pharmacodynamic effect, or 10 times the half-life of the drug, whichever is longer before providing a signed ICF.
* Donate blood more than 200 mL within 4 weeks, 400 mL within 12 weeks or 1000 mL within 52 weeks, respectively before providing a signed ICF.
* Donate plasma or platelet component within 2 weeks before providing a signed ICF.
* Use of any prescription or non-prescription medications including herbal remedies and vitamin/mineral/protein supplements, except for acetylsalicylic acid, within 7 days prior to IMPs dosing.
* Use of tobacco or nicotine containing products for 24 hours before each visit of screening or Day -1.
* Consumption of alcohol, xanthines, or grapefruit containing products for 24 hours before each visit of screening or Day -1.

Ages: 20 Years to 55 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 27 (Actual)
Dates: Start 2018-09-18 (Actual); Primary Completion 2018-10-20 (Actual); Study Completion 2018-10-23 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: General Manager, Study Director — Tanabe Pharma Corporation
Locations (1):
- Investigational site, Tokyo, Japan

REFERENCES:
- [Result] Shimizu H, Inoue S, Endo M, Nakamaru Y, Yoshida K, Natori T, Kakubari M, Akimoto M, Kondo K. A Randomized, Single-Blind, Placebo-Controlled, 3-Way Crossover Study to Evaluate the Effect of Therapeutic and Supratherapeutic Doses of Edaravone on QT/QTc Interval in Healthy Subjects. Clin Pharmacol Drug Dev. 2021 Jan;10(1):46-56. doi: 10.1002/cpdd.814. Epub 2020 Jun 15. PMID 32543120

RESULTS

PARTICIPANT FLOW:
Groups:
- Sequence 1 (Treatment A, Then Treatment C, Then Treatment B): Participants first received a single intravenous dose of Treatment A as 1-hour infusion. After 14day post treatment, they then received a single intravenous dose of Treatment C as 1-hour infusion. After 14day post treatment, they then received a single intravenous dose of Treatment B as 1-hour infusion. After 14day post treatment. (Treatment A=60mg of MCI-186, Treatment B=300mg of MCI-186, Treatment C=0.9% w/v saline)
- Sequence 2 (Treatment B, Then Treatment A, Then Treatment C): Participants first received a single intravenous dose of Treatment B as 1-hour infusion. After 14day post treatment, they then received a single intravenous dose of Treatment A as 1-hour infusion. After 14day post treatment, they then received a single intravenous dose of Treatment C as 1-hour infusion. After 14day post treatment. (Treatment A=60mg of MCI-186, Treatment B=300mg of MCI-186, Treatment C=0.9% w/v saline)
- Sequence 3 (Treatment C, Then Treatment B, Then Treatment A): Participants first received a single intravenous dose of Treatment C as 1-hour infusion. After 14day post treatment, they then received a single intravenous dose of Treatment B as 1-hour infusion. After 14day post treatment, they then received a single intravenous dose of Treatment A as 1-hour infusion. After 14day post treatment. (Treatment A=60mg of MCI-186, Treatment B=300mg of MCI-186, Treatment C=0.9% w/v saline)
Period: Overall Study
Arm/Group | Sequence 1 (Treatment A, Then Treatment C, Then Treatment B) | Sequence 2 (Treatment B, Then Treatment A, Then Treatment C) | Sequence 3 (Treatment C, Then Treatment B, Then Treatment A)
Started | 9 | 9 | 9
Completed | 8 | 8 | 9
Not Completed | 1 | 1 | 0
Not completed — Protocol Violation | 1 | 0 | 0
Not completed — Withdrawal by Subject | 0 | 1 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Sequence 1 (Treatment A, Then Treatment C, Then Treatment B) | Sequence 2 (Treatment B, Then Treatment A, Then Treatment C) | Sequence 3 (Treatment C, Then Treatment B, Then Treatment A) | Total
Number analyzed (Participants) | 9 | 9 | 9 | 27
Age, Continuous [Mean (Standard Deviation); unit: years] | 29.3 (9.8) | 28.7 (10.6) | 33.6 (9.8) | 30.5 (9.9)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0 | 0 | 0 | 0
  Male | 9 | 9 | 9 | 27
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0
  Asian | 9 | 9 | 9 | 27
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0
  Black or African American | 0 | 0 | 0 | 0
  White | 0 | 0 | 0 | 0
  More than one race | 0 | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0 | 0

OUTCOME MEASURES:

1. Primary Outcome: Change From Baseline in QTcF(ΔQTcF) With Placebo Adjustment (ΔΔQTcF) at Cmax of MCI-186
Description: The primary outcome endpoint was based on an analysis of the regression relationship between ΔQTcF and the concentration of MCI-186 at matching times post-dose, including adjustment for placebo treatments.
Time Frame: 45 min pre-dose to 24 h post-dose
Population: All participants who received 600mg, and 300mg of MCI-186 were included in the analysis. One participant on 300mg was not included due to meeting the exclusion criteria (Protocol Violation).
  Overall Number of Participants Analyzed was entered as the number at the time of calculation of Cmax.
Measure: Mean (90% Confidence Interval); unit: ms
Groups:
- MCI-186 60mg: A single dose of 60 mg MCI-186 over 60 min was intravenously administered.
- MCI-186 300mg: A single dose of 300 mg MCI-186 over 60 min was intravenously administered.
Arm/Group | MCI-186 60mg | MCI-186 300mg
Number analyzed (Participants) | 27 | 26
ms | -0.5 [-1.5 to 0.5] | 0.5 [-1.0 to 1.9]

2. Secondary Outcome: Change From Baseline of Heart Rate(HR) by Timepoint
Time Frame: Pre-dose to 24h post-dose
Population: All participants who received 600mg, 300mg, and placebo of MCI-186 were included in the analysis. One participant on 300mg , and one patient on placebo were not included due to meeting the exclusion criteria (Protocol Violation).
  One patient on placebo was not included due to withdrawal of the consent.
Measure: Mean (Standard Error); unit: beats per minute
Groups:
- Placebo: A single dose of 0.9% w/v saline over 60 min was intravenously administered.
Arm/Group | MCI-186 60mg | MCI-186 300mg | Placebo
Number analyzed (Participants) | 27 | 26 | 25
beats per minute
  30min | 0.2 (2.90) | -0.2 (2.47) | 0.1 (2.59)
  60min | 0.6 (3.21) | 1 (3.08) | 0.8 (3.02)
  75min | 1 (3.43) | 1.1 (3.14) | 1.1 (3.26)
  90min | 0.4 (3.17) | 1.8 (3.63) | 1.6 (3.81)
  105min | 0.6 (3.27) | 3.1 (3.55) | 1.8 (3.91)
  2hr | 1.7 (3.56) | 3.4 (3.24) | 3.4 (3.8)
  3hr | 1.8 (4.01) | 4 (3.69) | 2.6 (3.44)
  4hr | 2.1 (4.28) | 3.8 (4.22) | 3.1 (4.57)
  6hr | 7.6 (4.69) | 9.3 (5.18) | 9.1 (4.13)
  8hr | 8.1 (5.44) | 10.2 (6.26) | 10.3 (7.34)
  12hr | 7.1 (4.8) | 9.1 (6.77) | 7.4 (5.83)
  24hr | 1.1 (4.52) | 4.6 (6.9) | 2.7 (4.01)

3. Secondary Outcome: Change From Baseline of PR Interval by Timepoint
Time Frame: Pre-dose to 24h post-dose
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: msec
Arm/Group | MCI-186 60mg | MCI-186 300mg | Placebo
Number analyzed (Participants) | 27 | 26 | 25
msec
  30min | -0.4 (3.72) | 0 (6.14) | -1 (6.29)
  60min | -2.1 (3.74) | -0.3 (6.79) | -1.4 (5.93)
  75min | -2.2 (4.43) | -1.8 (5.53) | -2.5 (4.68)
  90min | -2.3 (4.29) | -2.4 (6.81) | -2.8 (4.91)
  105min | -1.1 (4.17) | -2.2 (7.91) | -3.1 (5.51)
  2hr | -2.8 (4.51) | -3.2 (7.96) | -2.3 (7.2)
  3hr | -4 (6.05) | -5.1 (7.34) | -1.7 (6.46)
  4hr | -4.6 (5.81) | -6.4 (7.6) | -3.4 (5.99)
  6hr | -4.2 (5.99) | -5.9 (8.36) | -5.3 (8.64)
  8hr | -7.3 (6.01) | -7.8 (8.58) | -7.9 (7.49)
  12h | -2.4 (7.96) | -5.5 (10.72) | -3.5 (9.46)
  24hr | 1.4 (6.87) | -1 (7.73) | -0.6 (7.16)

4. Secondary Outcome: Change From Baseline of QRS Interval by Timepoint
Time Frame: Pre-dose to 24h post-dose
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: msec
Arm/Group | MCI-186 60mg | MCI-186 300mg | Placebo
Number analyzed (Participants) | 27 | 26 | 25
msec
  30min | 3.4 (5.03) | 3.4 (3.53) | 3.4 (3.65)
  60min | 4.7 (3.54) | 5 (5.23) | 4.1 (3.95)
  75min | 4.1 (5.02) | 4.1 (3.86) | 3.6 (3.98)
  90min | 3.5 (3.61) | 3.5 (4.4) | 3.2 (4.13)
  105min | 3.2 (3.94) | 3.2 (3.64) | 2.9 (4.45)
  2hr | 1.4 (3.35) | 2.1 (4.62) | 1.9 (3.85)
  3hr | 0.2 (4.57) | -0.4 (4.47) | 0.1 (5.56)
  4hr | 0.7 (5.47) | -0.6 (6.06) | 1.4 (5.56)
  6hr | -7.3 (7.31) | -5.8 (7.42) | -4.8 (6.48)
  8hr | -6.4 (7.39) | -6.4 (6.63) | -5.5 (7.9)
  12hr | -6.4 (6.26) | -7 (7.86) | -4.2 (7.99)
  24hr | -6 (4.15) | -8 (5.13) | -5.6 (5.06)

5. Secondary Outcome: Change From Baseline of QTcF by Timepoint
Time Frame: Pre-dose to 24h post-dose
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: msec
Arm/Group | MCI-186 60mg | MCI-186 300mg | Placebo
Number analyzed (Participants) | 27 | 26 | 25
msec
  30min | 0.7 (1.91) | -1.8 (5.06) | 0.2 (1.94)
  60min | 0.2 (1.87) | -0.7 (3.62) | -0.1 (1.95)
  75min | -0.6 (1.83) | -1.1 (3.59) | -0.7 (2.92)
  90min | 0.1 (2.53) | -1.3 (4.15) | -0.9 (3.24)
  105min | -0.3 (2.7) | -1.3 (3.41) | -0.8 (2.53)
  2hr | -0.4 (3.28) | -2.1 (6.03) | -1.5 (3.31)
  3hr | 0.3 (3.27) | -2 (5.31) | -0.4 (2.42)
  4hr | 0.4 (3.08) | -2 (5.46) | -1 (2.38)
  6hr | 1.5 (3.17) | 3.5 (6.97) | 2.1 (4.05)
  8hr | 0.6 (3.39) | 0.3 (5.16) | 0.9 (5.32)
  12hr | 0.5 (3.99) | 0.4 (4.14) | 0.9 (3.33)
  24hr | 0 (3.82) | -0.7 (5.56) | -0.2 (2.9)

6. Secondary Outcome: Plasma Concentration of MCI-186
Time Frame: Pre-dose to 24h post-dose
Population: All participants who received 600mg, and 300mg of MCI-186 were included in the analysis. One participant on 300mg was not included due to meeting the exclusion criteria (Protocol Violation).
Measure: Mean (Standard Deviation); unit: ng/mL
Arm/Group | MCI-186 60mg | MCI-186 300mg
Number analyzed (Participants) | 27 | 26
ng/mL
  30min | 1039 (140.0) | 7393 (1770)
  60min | 791.3 (147.0) | 7412 (1968)
  75min | 454.4 (101.6) | 4864 (1606)
  90min | 308.3 (71.22) | 3522 (1235)
  105min | 227.6 (54.48) | 2578 (932.7)
  2hr | 176.1 (43.85) | 1990 (733.5)
  3hr | 83.60 (23.66) | 874.5 (326.8)
  4hr | 51.28 (15.49) | 512.7 (197.6)
  6hr | 20.39 (7.148) | 166.3 (69.70)
  8hr | 12.34 (4.689) | 89.91 (39.59)
  12hr | 6.522 (2.652) | 37.48 (16.83)
  24hr | 2.684 (1.547) | 10.65 (4.026)

7. Secondary Outcome: Pharmacokinetic(PK) Parameters - Area Under the Concentration Versus Time Curve From Time Zero to Infinity (AUC 0-inf) of MCI-186
Time Frame: Pre-dose to 24h post-dose
Population: as for outcome 6
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ng·h/mL
Arm/Group | MCI-186 60mg | MCI-186 300mg
Number analyzed (Participants) | 27 | 26
ng·h/mL | 1549.22 (20.5) | 12916.94 (33.3)

8. Secondary Outcome: PK Parameters - Maximum Plasma Concentration (Cmax) of MCI-186
Time Frame: Pre-dose to 24h post-dose
Population: as for outcome 6
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ng/mL
Arm/Group | MCI-186 60mg | MCI-186 300mg
Number analyzed (Participants) | 27 | 26
ng/mL | 1030 (14.1) | 7566 (25.1)

9. Secondary Outcome: Number of Participants With Adverse Events (AEs)
Time Frame: Day 1 to 9
Population: as for outcome 2
Measure: Count of Participants; unit: Participants
Arm/Group | MCI-186 60mg | MCI-186 300mg | Placebo
Number analyzed (Participants) | 27 | 26 | 25
Participants | 1 | 1 | 1

ADVERSE EVENTS:
Time Frame: up to 9 days
Description: All participants who received 600mg, 300mg, and placebo of MCI-186 were included in the analysis. One participant on 300mg , and one patient on placebo were not included due to meeting the exclusion criteria (Protocol Violation).
  One patient on placebo was not included due to withdrawal of the consent.
Arm/Group | MCI-186 60mg | MCI-186 300mg | Placebo
All-Cause Mortality (participants affected / at risk) | 0/27 | 0/26 | 0/25
Serious Adverse Events (participants affected / at risk) | 0/27 | 0/26 | 0/25
Other Adverse Events (participants affected / at risk) | 1/27 | 1/26 | 1/25
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | MCI-186 60mg (N=27) | MCI-186 300mg (N=26) | Placebo (N=25)
Gastroenteritis (Infections and infestations) | 0 | 1 | 0
Pharyngitis (Infections and infestations) | 1 | 0 | 0
Headache (Nervous system disorders) | 0 | 0 | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other

DOCUMENTS (2):
  • Study Protocol (2018-08-29): https://cdn.clinicaltrials.gov/large-docs/90/NCT04029090/Prot_000.pdf
  • Statistical Analysis Plan (2019-01-25): https://cdn.clinicaltrials.gov/large-docs/90/NCT04029090/SAP_001.pdf